CLINICAL TRIAL: NCT05004740
Title: Is COVID-19 Transmitted Through Human Milk? Implications for Breastfeeding and Human Milk Banking-Study 1c
Status: Completed | Type: Observational
Sponsor: Deborah O'Connor (Other)
Collaborators: University of Toronto (Other); Sinai Health System (Other)
Responsible Party: Sponsor-Investigator, Deborah O'Connor, Scientist, The Hospital for Sick Children
Organization: The Hospital for Sick Children (Other)
Other Study IDs: 39373-c
Record Dates: First submitted 2021-08-11; First posted 2021-08-13 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: COVID-19 Vaccine; Breastmilk

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lactating birthing persons delivering at Sinai Health System or from the general population
  Interventions: Other: Vaccinated Pregnant or Lactating persons

INTERVENTIONS:
Other: Vaccinated Pregnant or Lactating persons — vaccinated lactating persons from Sinai Health System or the general public

SUMMARY:
This will be a prospective observational study of lactating mothers who are planning to, have scheduled or have received vaccination against SARS-COV-2 (COVID-19 vaccine). Mothers may have delivered at Mount Sinai Hospital or may be from the general public recruited by social media or word of mouth. As the study participants will be lactating mothers, they will not be under the care of the investigators. Due to lack of information, we are unsure of an appropriate sample size but envision we will recruit at least 10 women each immunized with the approved mRNA vaccines (e.g. Pfizer-BioNTech and Moderna COVID-19 vaccines) and in the future at least two other vaccines (e.g. Oxford-AstraZeneca) as they are approved and become available. Milk samples will be analyzed for the presence of antibody to SARS-CoV-2 using the Anti-SARS-CoV-2 ELISA (IgG and IgA). These analyses will be conducted in the Department of Microbiology at Sinai Health following validation of the procedures in human milk.

ELIGIBILITY:
Inclusion Criteria:

* lactating birthing persons from the general public or Sinai Health System

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2021-01-17 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Number of participants with and timing of SARS-CoV-2 specific antibodies in breastmilk post-vaccination | Week prior to first dose of vaccination and until 4 weeks following the second dose of vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- Sinai Health System, Toronto, Ontario, Canada

REFERENCES:
- [Background] Ismail S, Unger S, Budylowski P, Poutanen S, Yau Y, Jenkins C, Anwer S, Christie-Holmes N, Kiss A, Mazzulli T, Johnstone J, McGeer A, Whittle W, Parvez B, Gray-Owen SD, Stone D, O'Connor DL. SARS-CoV-2 antibodies and their neutralizing capacity against live virus in human milk after COVID-19 infection and vaccination: prospective cohort studies. Am J Clin Nutr. 2024 Feb;119(2):485-495. doi: 10.1016/j.ajcnut.2023.10.008. Epub 2023 Dec 14. PMID 38309831